CLINICAL TRIAL: NCT05880602
Title: Clinical Trial of Nettle and Cranberry Capsules for Prevention of Urinary Tract Infection
Brief Title: Nettle and Cranberry Capsules for Prevention of Urinary Tract Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: Glory Kingdom Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS2-23025
Record Dates: First submitted 2023-05-19; First posted 2023-05-30 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Urinary Tract Infection
Keywords: Nettle; Cranberry; Prevention; Urinary Tract Infection; Recurrent Infection; Inflammation
MeSH Terms: conditions — Urinary Tract Infections; Reinfection; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Subjects will take two capsule of containing starch, twice a daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo(starch)
- Treatment (Experimental): Subjects will take two capsule of containing nettle and cranberry complex, twice a daily for 8 weeks.
  Interventions: Dietary Supplement: Nettle and Cranberry complex capsules

INTERVENTIONS:
Dietary Supplement: Nettle and Cranberry complex capsules — A specific capsule product, containing nettle and cranberry complex will be given to participants for oral intake for 8 weeks.
  Arms: Treatment
Dietary Supplement: Placebo(starch) — A specific capsule product, containing starch will be given to participants for oral intake for 8 weeks.
  Arms: Control

SUMMARY:
This study investigates whether the oral intake of a nettle and cranberry complex capsule may prevent recurrent urinary tract infection (rUTI). Participants will be aged between 30 - 75 years of age, with confirmed diagnosis of UTI status. The participants will be assessed for several parameters and asked to take 2 nettle and cranberry complex capsules twice daily for 8 weeks. The parameters will include international prostate symptoms score (IPSS), overactive bladder symptom score (OABSS), international consultation on incontinence questionnaire - overactive bladder (ICIQ-OAB), 3-day bladder diary (3dBD), and urine routine.

DETAILED DESCRIPTION:
Urinary tract infections (UTIs) are one of the most common bacterial infections affecting women. UTI occurs in 50-80% of women in the general population. About one in four women with one UTI episode will go on to develop frequent recurrences.

Recurrent urinary tract infection (rUTI) is defined as repeated UTI with a frequency of at least two episodes in the preceding six months or three episodes in the past year. rUTI has been regarded as a substantial global healthcare problem.

This investigation is a randomized, double-blind study. Subjects with confirmed diagnosis of rUTI are randomly assigned to control group or treatment group, and asked to orally intake 2 capsules of either placebo or nettle and cranberry complex capsules twice daily. Participants will be assessed for parameters, including international prostate symptoms score (IPSS) (male only), overactive bladder symptom score (OABSS), international consultation on incontinence questionnaire - overactive bladder (ICIQ-OAB), 3-day bladder diary (3dBD) and urine routine. The assessments are conducted at baseline, 4 weeks, and 8 weeks after the oral intake period. The parameters are used to compare and evaluate whether the nettle and cranberry complex capsule can prevention rUTI.

ELIGIBILITY:
Inclusion Criteria:

* aged between 30 and 75 years
* at least two episodes in 6 months, or at least three episodes of a UTI in 12 months.

Exclusion Criteria:

* pregnancy women
* diabetes
* History of anatomical urogenital anomalies, urogenital tract surgery
* History of acute or chronic renal failure, nephrolithiasis
* History of intestinal diseases causing malabsorption
* Anticoagulant medication in the last month
* immunocompromise
* Known allergy or intolerance to cranberry

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
UTI-free duration in 8 weeks | on baseline and 8 weeks
  Comparing the number of days from the beginning of the study to the first recurrence of UTI, and the number of days from each recurrence to the next recurrence between different treatment groups.
UTI recurrent incidence in 8 weeks | 8 weeks
  UTI episodes during 8 weeks treatment for each subject

SECONDARY OUTCOMES:
International Prostate Symptom Score (IPSS) Change from Baseline | on baseline,4 weeks and 8 weeks
  The IPSS questionnaire is a tool commonly used to assess the severity of LUTS, and to monitor the progress of the symptoms during treatment. Score range is 0-35, with higher scores indicating increasing symptom severity.
Overactive Bladder Symptom Score (OABSS) Change from Baseline | on baseline,4 weeks and 8 weeks
  OABSS is a valid self-assessment questionnaire, with four questions set according to OAB syndrome to determine the severity of OAB, which includes daytime and nighttime urination frequency, urgency, and urge incontinence. Score range is 0-15, with higher scores indicating increasing symptom severity.
International Consultation on Incontinence Questionnaire Overactive Bladder Score (ICIQ-OAB) Change from Baseline | on baseline,4 weeks, and 8 weeks
  Assessment of quality of life related to the impact of overactive bladder symptoms on daily activities.
  Assessment of quality of life related to the impact of overactive bladder symptoms on daily activities Assessment of quality of life related to the impact of overactive bladder symptoms on daily activities.
Bladder diary | on baseline,4 weeks, and 8 weeks
  Assessment of number of voids, number of leakages, and post void residual.

CONTACTS AND LOCATIONS:
Overall Officials: David Pei-Cheng Lin, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Stamm WE, Norrby SR. Urinary tract infections: disease panorama and challenges. J Infect Dis. 2001 Mar 1;183 Suppl 1:S1-4. doi: 10.1086/318850. No abstract available. PMID 11171002
- [Background] Harding GK, Ronald AR. The management of urinary infections: what have we learned in the past decade? Int J Antimicrob Agents. 1994 Jun;4(2):83-8. doi: 10.1016/0924-8579(94)90038-8. PMID 18611593
- [Background] Sivick KE, Mobley HL. Waging war against uropathogenic Escherichia coli: winning back the urinary tract. Infect Immun. 2010 Feb;78(2):568-85. doi: 10.1128/IAI.01000-09. Epub 2009 Nov 16. PMID 19917708
- [Background] Foxman B, Barlow R, D'Arcy H, Gillespie B, Sobel JD. Urinary tract infection: self-reported incidence and associated costs. Ann Epidemiol. 2000 Nov;10(8):509-15. doi: 10.1016/s1047-2797(00)00072-7. PMID 11118930
- [Background] Sihra N, Goodman A, Zakri R, Sahai A, Malde S. Nonantibiotic prevention and management of recurrent urinary tract infection. Nat Rev Urol. 2018 Dec;15(12):750-776. doi: 10.1038/s41585-018-0106-x. PMID 30361493
- [Background] Kwok M, McGeorge S, Mayer-Coverdale J, Graves B, Paterson DL, Harris PNA, Esler R, Dowling C, Britton S, Roberts MJ. Guideline of guidelines: management of recurrent urinary tract infections in women. BJU Int. 2022 Nov;130 Suppl 3(Suppl 3):11-22. doi: 10.1111/bju.15756. Epub 2022 May 17. PMID 35579121
- [Background] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Background] Guay DR. Cranberry and urinary tract infections. Drugs. 2009;69(7):775-807. doi: 10.2165/00003495-200969070-00002. PMID 19441868
- [Background] Scholes D, Hooton TM, Roberts PL, Stapleton AE, Gupta K, Stamm WE. Risk factors for recurrent urinary tract infection in young women. J Infect Dis. 2000 Oct;182(4):1177-82. doi: 10.1086/315827. Epub 2000 Aug 31. PMID 10979915
- [Background] Wan X, Wu C, Xu D, Huang L, Wang K. Toileting behaviours and lower urinary tract symptoms among female nurses: A cross-sectional questionnaire survey. Int J Nurs Stud. 2017 Jan;65:1-7. doi: 10.1016/j.ijnurstu.2016.10.005. Epub 2016 Oct 21. PMID 28027949